CLINICAL TRIAL: NCT05230901
Title: Effect of Antifibrotic Therapy on Regression of Myocardial Fibrosis After Transcatheter Aortic Valve Implantation (TAVI) in Aortic Stenosis Patients With High Fibrotic Burden
Acronym: Reduce-MFA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Karsten Gavenis, Clinical Study Management on behalf of the Principal Investigator, University Medical Center Goettingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02717
Record Dates: First submitted 2022-01-12; First posted 2022-02-09 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Aortic Stenosis, Severe
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Standard of Care; Spironolactone; Dihydralazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): Patients with CMR-derived ECV% levels ≥25.9% will receive Standard of care
  Interventions: Other: Standard of Care
- Spironolactone (Experimental): Patients with CMR-derived ECV% levels ≥25.9% will receive Standard of care + Spironolactone (25 mg/d, p.o.)
  Interventions: Other: Standard of Care; Drug: Spironolactone 25mg
- Spironolactone + Dihydralazine (Experimental): Patients with CMR-derived ECV% levels ≥25.9% will receive Standard of care + Spironolactone (25 mg/d, p.o.) + Dihydralazine (2x12.5 mg/d p.o. in slow acethylators, and 2x25mg / d p.o. in fast acethylators, confirmed by genetic testing)
  Interventions: Other: Standard of Care; Drug: Spironolactone 25mg; Drug: Dihydralazine

INTERVENTIONS:
Other: Standard of Care — Patients with CMR-derived ECV% levels ≥25.9% will be treated with standard of care according to current guidelines (Control group).
Drug: Spironolactone 25mg — Patients with CMR-derived ECV% levels ≥25.9% in Arm "Spironolactone" will receive spironolactone 25 mg/d in addition to standard of care medication .
  Arms: Spironolactone; Spironolactone + Dihydralazine
Drug: Dihydralazine — Patients with CMR-derived ECV% levels ≥25.9% in arm "Spironolactone + Dihydralazine" will receive spironolactone 25 mg/d + dihydralazine (2x12.5 mg/d p.o. in slow acethylators, and 2x25mg/d p.o. in fast acethylators, confirmed by genetic testing)
  Arms: Spironolactone + Dihydralazine

SUMMARY:
The aim of the study is to evaluate the effect of antifibrotic therapy on regression of myocardial fibrosis after TAVI in patients with baseline high fibrotic burden. Therefore, patients will be treated with Spironolactone in addition to standard of care, Spioronolactone + Dihydralazine in addition to standard of care or according to standard of care alone without any study medication. First, differences between patients in the control arm and patients randomized to anti-fibrotic therapy will be analyzed. The second analysis will determine, whether dihydralazine medication in addition to spironolactone is able to increase a potential antifibrotic effect. Myocardial fibrosis will be assessed by cardiac magnetic resonance imaging (CMR) before TAVI and 1 year after. Quantification of potentially irreversible replacement fibrosis will be carried out by late gadolinium enhancement (LGE), and quantification of the potentially reversible diffuse interstitial fibrosis will be performed by measurement of the extracellular volume fraction (ECV), thereby deriving matrix volume and cell volume.

ELIGIBILITY:
Inclusion Criteria:

* Male, female age ≥ 60
* Diagnosis of severe symptomatic aortic stenosis
* Transcatheter aortic valve implantation (TAVI) scheduled
* Written informed consent

Exclusion Criteria:

* 1. Pre-existing dilative or ischemic heart disease with EF<35% and guideline indication for spironolactone
* Patient on current medication with spironolactone, eplerenone, or dihydralazine
* Presence of coexistent myocardial pathology such as cardiac amyloidosis, hypertrophic cardiomyopathy, or myocarditis
* Presence of coexistent severe aortic regurgitation or severe mitral stenosis
* Previous surgical valve replacement or repair
* Pacemaker or ICD implanted
* Renal impairment (serum creatinine > 1,8 mg/dl and/ or GFR < 30 ml/min/1,73 m² BSA)
* Significant hypotension (blood pressure < 90 mm Hg systolic and/or < 50 mm Hg diastolic
* Serum potassium > 5,1 mmol/l
* Contraindications for Spironolactone (anuria, acute renal failure, serum creatinine > 1.8 mg/dl, hyperkalemia, pregnancy)
* Contraindications for Dihydralazine (known allergy or hypersensitivity, systemic lupus erythematodes, adrenocortical disorders)
* Known active malignant disease with life expectancy < 1 year
* Women with child-bearing potential
* Simultaneous participation (including a waiting period of 4 weeks) in other interventional clinical trials
* Patient without legal capacity who is unable to understand the nature, significance and consequences of the trial
* Person who is in a relationship of dependence/employment with the sponsor or the investigator

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Extracellular volume (ECV)-derived matrix volume (measured by CMR) | 12 months
  Differences between treatment groups in reduction of extracellular volume (ECV)- derived matrix volume (measured by CMR) after 12 months

SECONDARY OUTCOMES:
Left ventricular ejection fraction | 12 months
  Differences in recovery of left ventricular ejection fraction (EF) in % (measured by CMR) after 12 months
Global longitudinal strain | 12 months
  Differences in recovery of global longitudinal strain (GLS) in % (measured by CMR) after 12 months
diastolic function | 12 months
  Differences in recovery of diastolic function (measured by CMR) after 12 months
Left ventricular myocardial tissue volumes | 12 months
  Differences in reduction of left ventricular myocardial tissue volumes (measured by CMR) after 12 months
Left ventricular blood volumes | 12 months
  Differences in reduction of left ventricular blood volumes (measured by CMR) after 12 months
Kansas City Cardiomyopathy Questionnaire | 12 months
  Differences in quality of life changes according to 23-items Kansas City Cardiomyopathy Questionnaire (KCCQ) after 12 months
NYHA status | 12 months
  Differences in NYHA status after 12 months
6min-walking test distance (6MWT) | 12 months
  Differences in 6min-walking test distance (6MWT; in m) after 12 months
NT-proBNP-levels | 12 months
  Differences in NT-proBNP-levels (in pg/ml) after 12 months
Heart failure hospitalizations | 12 months
  Rate of Heart failure hospitalizations within 12 months
Total mortality | 12 months
  Rate of total mortality within 12 months
Cardiovascular mortality | 12 months
  Rate of Cardiovascular mortality within 12 months
Biomarker Procollagen type I carboxy-terminal propeptide (PICP) | 12 months
  Measurement of PICP in ng/ml
Biomarker Procollagen III N-terminal propeptid (PIIINP) | 12 months
  Measurement of PIIINP in ng/ml
Ratio of Increased collagen degradation (CITP) vs. matrix metalloproteinase-1 (MMP-1) | 12 months
  Measurement of CITP (in ng/l) and MMP-1 (in ng/ml)
Methylation of Iroquois Homeobox 3 (IRX3) | 12 months
  Measurement of Methylation of IRX3 in %
Methylation of rfGAP With Coiled-Coil, Ankyrin Repeat And PH Domains 3 (ACAP3) | 12 months
  Measurement of Methylation of ACAP3 in %
Methylation of Growth Arrest And DNA Damage Inducible Gamma (GADD45G) | 12 months
  Measurement of Methylation of GADD45G in %
Methylation of Chordin (CHRD) | 12 months
  Measurement of Methylation of CHRD in %
Methylation of Klotho | 12 months
  Measurement of Methylation of Klotho in %
Methylation of RAS Protein Activator Like 1 (RASAL1) | 12 months
  Measurement of Methylation of RASAL1 in %
Methylation of ATPase Sarcoplasmic/Endoplasmic Reticulum Ca2+ Transporting 2 (ATP2A2) | 12 months
  Measurement of Methylation of ATP2A2 in %
Methylation of B9 Domain Containing 1 (B9D1) | 12 months
  Measurement of Methylation of B9D1 in %
Methylation of Bone Morphogenetic Protein 7 (BMP7) | 12 months
  Measurement of Methylation of BMP7 in %
Methylation of Latency associated peptide (LAP) | 12 months
  Measurement of Methylation of LAP in %
Serum creatinine | 12 months
  Change in serum creatinine (in mg/dl) after 12 months
Cystatin c | 12 months
  Change in cystatin c (in mg/l) after 12 months
Phosphate | 12 months
  Change in phosphate (in mmol/l) after 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Göttingen, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No